CLINICAL TRIAL: NCT06988930
Title: To Compare the Clinical Efficacy of Arthroscopic Lateral Retinacular Release and Exercise Therapy in the Treatment of Lateral Patellar Crush Syndrome
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2024181
Record Dates: First submitted 2025-04-07; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: Lateral Patellar Syndrome
Keywords: lateral patellar compression syndrome; lateral retinacular release of the patella; patellofemoral joint rehabilitation; prospective cohort study; kinesitherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group：arthroscopic surgery (Experimental): The patients with lateral patellar extrusion were treated with arthroscopic minimally invasive surgery.
  Interventions: Diagnostic Test: Control group
- Conservative rehabilitation training group (Active Comparator): The patients in this group were treated with exercise therapy
  Interventions: Diagnostic Test: Control group

INTERVENTIONS:
Diagnostic Test: Control group — The non-operation group was treated with rehabilitation therapy for 6 weeks, and the operation group was treated with arthroscopic surgery and the pathological tissue of cartilage and subchondral bone was taken. Assessment was performed at three months, one year, and two years after treatment and recorded in the database.

SUMMARY:
One hundred patients with lateral patellar compression syndrome (LPCS) were recruited and divided into two groups: arthroscopic treatment group and rehabilitation conservative treatment group. A 2-year prospective cohort study was then conducted. The subjective scores of 5 scales and 3 objective indexes were used to evaluate the recovery of knee joint function after different treatment methods, and to further clarify the medium and long-term therapeutic effects of different treatment methods on LPCS patients.

DETAILED DESCRIPTION:
Lateral patellar over-compression syndrome is a musculoskeletal disease characterized by increased pressure on the lateral patellofemoral joint, which is caused by long-term tilting of the patella, adaptive contraction of the lateral retinaculum and long-term stress imbalance of the medial and lateral articular surfaces. The main clinical manifestations are patellofemoral joint pain, abnormal patellar trajectory and articular cartilage injury. At present, the prevalence of anterior knee pain is as high as 8. 5% ~ 17. 0%, and female is higher than male. LPCS has become one of the main causes of anterior knee pain . There are many methods for the treatment of LPCS, some of which are still controversial. At present, the gold standard for the treatment of LPCS has not been determined.

In the clinical practice of the Institute of Sports Medicine and the previous scientific research of our group, we found that a considerable number of patients, after arthroscopic patella molding, lateral retinaculum release and joint cleaning, their pain was obviously relieved, the patella trajectory almost returned to normal, and the knee joint symptoms were well improved and returned to normal life.

Both arthroscopic surgery and conservative rehabilitation can be used to treat LPCS, but it has not been proved that the functional improvement and symptom improvement rate of the two treatment methods are better in the medium and long term follow-up. Based on the above background, this study will conduct a prospective cohort study, and plan to recruit 100 patients and divide them into two groups, namely the arthroscopic group and the conservative treatment group, for a 2-year follow-up. The patients' subjective scores of 5 scales and 3 objective indicators were used to evaluate the recovery of knee function after different treatment methods, and to further clarify the medium and long-term therapeutic effects of different treatment methods on patients with LPCS, in order to provide guidance and reference for the clinical treatment of LPCS.

ELIGIBILITY:
Inclusion Criteria:

* ① Meet the diagnostic criteria of LPCS; ② Complete imaging data; ③ agree that the follow-up time should be at least 1 Years; ④ Those who are willing to conduct regular rehabilitation training can cooperate to complete the experiment by signing the informed consent.

Exclusion Criteria:

* ① Complicated with severe heart, brain, kidney and other organ dysfunction;② Combined with patellar instability, patellar dislocation or others Severe knee joint disease and injury; ③ The previous history of joint infection, joint tuberculosis or osteomyelitis, or the lower extremity in 6 A history of surgery within the last month and previous knee surgery; ④ Infection, cancer, pregnancy and mental disorders Those with special conditions. ⑤ patients with mental illness or cognitive impairment, unable to study and participate in rehabilitation training; ⑥ not Informed consent was obtained.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patellar axial X-ray | Before the intervention、3 months after the intervention and 1 year after the intervention
  The degree of deviation of the patella was evaluated mainly by X-ray measurement

SECONDARY OUTCOMES:
Visual Analogue Score | Before the intervention、3 months after the intervention and 1 year after the intervention
  The Visual Analog Scale (VAS) is a tool used to assess pain or other subjective sensations. It is typically represented by a line segment, with one end indicating no pain or symptoms and the other end indicating the most severe pain or symptoms. In clinical research, the VAS is commonly used to evaluate the level of pain experienced by patients. Patients mark their pain level on a line segment that is marked from 0 to 10 , where 0 represents no pain and 10 represents the most severe pain.
Kujala score | Before the intervention、3 months after the intervention and 1 year after the intervention
  The Kujala score is a system used to assess knee function. It quantifies pain, functional impairment, muscle strength, range of motion, swelling, and crepitus in the knee joint through a series of questions and examinations, thereby evaluating the overall condition of the knee. The score ranges from 0 to 100, with 100 being the highest possible score. A higher score indicates better knee function and less pain and functional impairment. Conversely, a lower score indicates severe knee dysfunction and significant pain and impairment. It is widely used in the diagnosis of knee-related diseases, evaluation of treatment outcomes, and rehabilitation guidance.
Lysholm knee score scale | Before the intervention、3 months after the intervention and 1 year after the intervention
  The Lysholm knee score scale is mainly used to assess the functional recovery of the knee joint after injury or surgery and can also be applied in clinical research of knee joint diseases. It focuses on the patient's subjective feelings and ability to perform daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes